CLINICAL TRIAL: NCT03191760
Title: Open Trial of Behavioral Activation and Social Engagement (BASE) for Posttraumatic Stress Disorder (PTSD)
Acronym: PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tracy Simpson, Clinician Investigator, VA Puget Sound Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00975
Record Dates: First submitted 2017-06-09; First posted 2017-06-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Social Support; Primary Care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Activation and Social Engagement (Experimental): Participants will attend 6 in-person or phone-mediated therapy sessions lasting approximately 45 minutes per session, held in Primary Care settings. Content of therapy sessions includes education about PTSD symptoms, discussion of the role of avoidance in maintaining PTSD symptoms, self-monitoring homework to identify links between activity level and emotions, and homework designed to increase engagement in valued activities, with a focus on increasing social contact and support. If relevant, participants will be instructed in basic communication skills, social skills, and relaxation skills. We have modified the standard Behavioral Activation intervention by reducing the number and length of sessions to accommodate the Primary Care setting. In addition, there will be a stronger emphasis on social engagement in BASE then in standard BA and social contact and support will be addressed during each treatment session.
  Interventions: Behavioral: Behavioral Activation

INTERVENTIONS:
Behavioral: Behavioral Activation — Participants will be asked to attend 6 in-person or phone-mediated therapy sessions lasting approximately 45 minutes per session, to be held in Primary Care settings. Content of therapy sessions includes education about PTSD symptoms, discussion of the role of avoidance in maintaining PTSD symptoms, self-monitoring homework to identify links between activity level and emotions, and homework designed to increase engagement in valued activities, with a focus on increasing social contact and support. If relevant, participants will be instructed in basic communication skills, social skills, and relaxation skills.

SUMMARY:
The purpose of the study is to see if "Behavioral Activation and Social Engagement for PTSD" (BASE for PTSD), an individual therapy for PTSD, will help Veterans with PTSD 1) through improved understanding of how PTSD affects them, 2) by reducing ways in which they avoid meaningful activity due to PTSD, 3) by enabling them to do more of the things they really care about, and 4) by improving, strengthening, and building up their social supports.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a mental health condition that some people develop following exposure to a traumatic event. PTSD often results in a reduction in feelings of connection to other people and changes in views about others, as well as reduced participation in valued activities. Many veterans with PTSD do not seek treatment offered in specialty mental health settings and may forgo treatment of any kind.

This study is an open-trial format (no comparison condition) of U.S. military veterans who will participate in a brief psychotherapy treatment for PTSD offered in a Primary Care setting. This is a pilot trial to see if the treatment is effective at reducing symptoms of PTSD and increasing feelings of social support, and an exploratory aim is to see if veterans engage in additional treatment after completing this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who:

  1. are currently enrolled in either of the Primary Care Clinics (including Women's Clinic) or Primary Care Mental Health Integration clinic at VA Puget Sound Health Care System - Seattle Division
  2. meet criteria for clinical or subclinical PTSD
  3. are willing to have therapy sessions audiotaped for the purposes of supervision
  4. plan to live in the Seattle area for 6 months following entry into the study

Exclusion Criteria:

* Veterans who:

  1. exhibit the presence of severe mental illness diagnosis (e.g., active psychosis and/or uncontrolled bipolar disorder)
  2. have been a psychiatric in-patient admission in the past 30 days
  3. have had a suicide attempt in the last 60 days
  4. have had a plan or intent to harm self or others in the last 30 days
  5. have a behavioral flag in their medical record
  6. have had a psychiatric medication dosing or receipt that has changed in the last 30 days
  7. are unwilling to provide at least 1 collateral contact
  8. have impaired decision making capacity (as measured by evidence in the Computerized Patient Record System record of moderate-severe Traumatic Brain Injury, uncontrolled psychosis, dementia, communication flag, or by clinical judgment in speaking with the participant
  9. are prisoners
  10. are illiterate or have limited or no English proficiency
  11. are terminally ill
  12. are currently participating in Cognitive Processing Therapy (CPT) or Prolonged Exposure Therapy (PE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist-Military Version | baseline to 4 weeks, 4 weeks to 8 weeks, 8 weeks to 12 weeks
  Change in PTSD symptoms
Medical Outcomes Study Social Support Survey Form and Social Connectedness Scale - Revised | baseline to 4 weeks, 4 weeks to 8 weeks, 8 weeks to 12 weeks
  Change in social support
Patient Health Questionnaire-9 | baseline to 4 weeks, 4 weeks to 8 weeks, 8 weeks to 12 weeks
  Change in Depression symptoms
Network Orientation Scale | baseline to 4 weeks, 4 weeks to 8 weeks, 8 weeks to 12 weeks
  Change in social network orientation
Behavioral Activation for Depression Scale | baseline to 4 weeks, 4 weeks to 8 weeks, 8 weeks to 12 weeks
  Change in activity level

SECONDARY OUTCOMES:
Qualitative assessment | 12 weeks
  Participants' reactions to the treatment will be gathered in qualitative interviews assessing treatment experience, perceptions of treatment focus, engagement with valued activities, social support, therapeutic relationship
Additional treatment engagement | 16 weeks
  measured via medical record review
Brief COPE | baseline to 4 weeks, 4 weeks to 8 weeks, 8 weeks to 12 weeks
  Change in coping strategies
Social Connectedness Scale - Revised (SCS-R) | baseline to 4 weeks, 4 weeks to 8 weeks, 8 weeks to 12 weeks
  Change in the level of interpersonal closeness related to participants' social environment and the degree of difficulty experienced by participants in sustaining the sense of closeness

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Simpson, PhD, Principal Investigator — Research Scientist
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT03191760/ICF_000.pdf